CLINICAL TRIAL: NCT00746837
Title: A Phase I Study to Assess Absolute Bioavailability of AZD5672 at Steady-state in Healthy Volunteers
Brief Title: AZD5672 Absolute Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Layton, MD, PhD, Medical Science Director, AstraZeneca R&D Alderely Park
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: D1710C00018; EudraCt nr 2008-003933-25
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers
Keywords: AZD5672
MeSH Terms: interventions — N-(1-(3-(3,5-difluorophenyl)-3-(4-methanesulfonylphenyl)propyl)piperidin-4-yl)-N-ethyl-2-(4-methanesulfonylphenyl)acetamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Single ascending IV dose, 3 treatment periods separated by a minimum 14 day washout between doses
  Interventions: Drug: AZD5672
- 2 (Experimental): 2 cohorts single IV dose + multiple oral dose period separated by a minimum of 14 days washout between IV and oral dose
  Interventions: Drug: AZD5672

INTERVENTIONS:
Drug: AZD5672 — single IV doses starting at 7 mg, subsequent doses to be confirmed following review of PK and safety data after each treatment period
Drug: AZD5672 — 50 mg od, 12 days
  Arms: 2
Drug: AZD5672 — 150mg od, 12 days
  Arms: 2

SUMMARY:
The purpose of the study is to estimate the absolute bioavailability at steady state of 2 doses of AZD5672 (50 mg and 150 mg administered orally once daily)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Females should not be of childbearing potential
* Clinically normal physical and laboratory findings as judged by the investigator, including negative test results for drug-of-abuse, alcohol and cotinine at the Screening Visit and/or admission (Day -1) of each study period, and negative test results

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subject's ability to participate
* Unsuitable venous access for intravenous studies
* Participation in a clinical study involving an investigational product within 5 half-lives of active moieties of the last dose of investigational product or 3 months prior to first dosing (whichever is longer).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during study periods

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, MD, PhD, Study Director — AstraZeneca R&D, Charnwood, UK; Tania Hugo, Principal Investigator — PAREXEL Clinical Pharmacology Research Unit
Locations (1):
- Research Site, Harrow, London, United Kingdom